CLINICAL TRIAL: NCT05032235
Title: A Multi-centre, Open-label and Parallel-control Study to Investigate the Pharmacokinetics of Fluzoparib in Healthy Subjects and Those With Impaired Kidney Function
Brief Title: Safety and Pharmacokinetics of Fluzoparib in Healthy Subjects and Those With Impaired Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SHR3162-I-119
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — fluzoparib

STUDY DESIGN:
Intervention Model Description: Single dose of oral administration of Fluzoparib
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental)
  Interventions: Drug: Fluzoparib
- Group B (Experimental)
  Interventions: Drug: Fluzoparib
- Group C (Experimental)
  Interventions: Drug: Fluzoparib

INTERVENTIONS:
Drug: Fluzoparib — Normal Renal Function:A single oral dose of Fluzoparib will be administered.
  Arms: Group A
Drug: Fluzoparib — Mild Renal Impairment:A single oral dose of Fluzoparib will be administered.
  Arms: Group B
Drug: Fluzoparib — Moderate Renal Impairment:A single oral dose of Fluzoparib will be administered.
  Arms: Group C

SUMMARY:
The primary objective is to evaluate pharmacokinetics of Fluzoparib and its main metabolite in subjects with impaired kidney function in comparison with healthy subjects, to develop dose recommendations for patients with renal impairment.

The secondary objective is to evaluate the safety of Fluzoparib in subjects with mild and moderate renal impairment and in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion Criteria for subjects with impaired kidney function:

1. Sign the informed consent before the trial, and fully understand the content, process, and possible adverse reactions of the trial;
2. Male or female subjects aged 18 to 70 (including 18 and 70);
3. Body mass index (BMI) ranges from 18 kg/m2 to 28 kg/m2 (including 18 and 28);
4. The glomerular filtration rate should meet the following criteria (GFR, mL/min):Subjects with mild renal impairment (CKD2): 60-89 mL/min (including 60-89);Subjects with moderate renal impairment (CKD3): 30-59 mL/min (including 30-59 ends);
5. Renal function should be stable, and the GFR results should be tested twice before administration (at least 3 days apart) within the same CKD stage.

Inclusion Criteria for subjects with normal kidney function:

1. Sign the informed consent before the trial and fully understand the content, process, and possible adverse reactions of the trial;
2. Male or female subjects aged 18 to 70 (including 18 and 70);
3. Body mass index (BMI) ranges from 18 kg/m2 to 28 kg/m2 (including 18 and 28);
4. Glomerular filtration rate (GFR) ≥90 mL/min.

Exclusion Criteria:

-

Exclusion Criteria for subjects with impaired kidney function:

1. History of kidney transplant;
2. Need Renal dialysis during the study;
3. Urinary incontinence or anuria;
4. Clinically significant heart disease, including but not limited to: congestive heart failure, symptomatic coronary artery disease, myocardial infarction, QTcF≥470 ms (female) or QTcF≥450 ms (male) within 12 months before the start of treatment;
5. Received any investigational drug within 3 months before the study started;
6. Taking any drugs which can affect the metabolic enzyme CYP3A within 14 days before the study started;
7. Smokers and alcoholics, or those screened positive for alcohol;
8. History of drug use, or drug abuse screening positive.

Exclusion Criteria for subjects with normal kidney function:

1. History of kidney transplant;
2. Clinically significant heart disease, including but not limited to: congestive heart failure, symptomatic coronary artery disease, myocardial infarction, QTcF≥470 ms (female) or QTcF≥450 ms (male) within 12 months before the start of treatment;
3. Received any investigational drug within 3 months before the study started;
4. Taking any drugs which can affect the metabolic enzyme CYP3A within 14 days before the study started;
5. Smokers and alcoholics, or those screened positive for alcohol;
6. History of drug use, or drug abuse screening positive.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters of Fluzoparib: Cmax | 96 hours post dose
Pharmacokinetics parameters of Fluzoparib: AUC0-t | 96 hours post dose
Pharmacokinetics parameters of Fluzoparib: AUC0-∞ (if available) | 96 hours post dose
Pharmacokinetics parameters of main metabolite (SHR165202) of Fluzoparib: Cmax | 96 hours post dose
Pharmacokinetics parameters of main metabolite (SHR165202) of Fluzoparib: AUC0-t | 96 hours post dose
Pharmacokinetics parameters of main metabolite (SHR165202) of Fluzoparib: AUC0-∞ (if available) | 96 hours post dose

SECONDARY OUTCOMES:
Other pharmacokinetics parameters of Fluzoparib: Tmax | 96 hours post dose
Other pharmacokinetics parameters of main metabolite (SHR165202) of Fluzoparib: Tmax | 96 hours post dose
Plasma protein binding rate of Fluzoparib | Day 01 post dose
Plasma protein binding rate of main metabolite (SHR165202) of Fluzoparib | Day 01 post dose
The incidence and severity of adverse events/serious adverse events (based on NCI-CTCAE 5.0) | 19 days

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of Chongqing medical university, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided